CLINICAL TRIAL: NCT01193205
Title: Evaluating the Effectiveness of Dialectical Behaviour Skills Training for Suicidality in Borderline Personality Disorder
Brief Title: 20 Weeks DBT Group Skills Training Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Shelley McMain, Head, Borderline Personality Disorder Clinic, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050/2010
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Skills Training; Dialectical Behavior Therapy; Suicidal and parasuicidal behavior
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20 weeks skills group (Experimental): Participants receive 20 weeks of Dialectical Behaviour Therapy Skills training, covering 5 modules: mindfulness, interpersonal effectiveness, emotional regulation, distress tolerance, dialectics.
  Interventions: Behavioral: Skills Training
- Waitlist (No Intervention): Participants on the waitlist condition will be assessed at baseline and symptoms monitored at 10 weeks, 20 weeks and 8 months following baseline assessment. They will then be offered the active treatment.

INTERVENTIONS:
Behavioral: Skills Training — 20 weeks of Dialectical Behaviour Therapy Skills Training
  Arms: 20 weeks skills group

SUMMARY:
The aim of this study is to evaluate the effectiveness of a 20-week Dialectical Behaviour Therapy (DBT) skills training group for the treatment of chronic suicidal and non-suicidal self-injurious (NSSI) behaviours in individuals diagnosed with borderline personality disorder (BPD). Previous research has established the effectiveness of a one year comprehensive, combined individual and group DBT treatment. However, in practice, DBT is often offered in a skills only group format. This study will consist of a randomized, controlled trial designed to evaluate the effectiveness of DBT compared to a wait list control. 84 participants will be randomized to the 20-week DBT group or the wait-list and the following outcomes will be assessed:

1. frequency of suicidal and NSSI behaviours
2. symptom distress
3. impulsivity
4. treatment retention
5. skill acquisition and
6. social functioning

Assessments will occur at pre-treatment, 10 weeks, 20 weeks and 3 months post treatment. The following main hypotheses will be examined: (1) Patients in the DBT skills group condition will have superior outcomes to patients on the treatment as usual wait list control in areas targeted by the treatment: frequency of suicidal and NSSI behaviours, emergency room visits, psychiatric hospital admissions, impulsivity, and knowledge and use of behavioral skills, general symptoms. The group receiving DBT will have superior outcomes at post treatment and these outcomes will be maintained during the three month post-treatment follow-up.

DETAILED DESCRIPTION:
The study will consist of a single-blind, two-arm randomized controlled trial designed to evaluate the effectiveness of DBT skills group offered as an adjunct to treatment as usual compared to a wait list control plus treatment as usual. The continuation of treatment as usual in both arms is permitted for two reasons. First, it would be unethical to assign suicidal patients to a wait list condition that prohibited involvement in ongoing treatment. Second, the proposed design enables us to address the question of the additive effect of the DBT skills group intervention. Subjects will be randomized to receive 20 weeks of DBT group skills training plus treatment as usual, or to a wait list control plus treatment as usual. Clinical effectiveness outcomes will be assessed at baseline, at 10 weeks, at 20 weeks and at 8 months follow-up. DBT skills training is a manualized intervention developed by Linehan (1993). Key skills from the modules described in Miller, Rathus, and Linehan (2006) will serve as the basis of the DBT skills group, delivered in a psychoeducational format over the course of weekly two-hour sessions. The skills group covers five modules: mindfulness, emotion regulation, distress tolerance, interpersonal effectiveness, and dialectics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DSM-IV Borderline Personality Disorder
* 18-60 years of age
* have had two suicidal or non-suicidal self-injurious behaviours in the past five years with one occurring in the past ten weeks
* be literate in English
* provide informed consent to participate in the study.

Exclusion Criteria:

* not meet DSM-IV criteria for a psychotic disorder, bipolar disorder or, dementia
* not have evidence of an organic brain syndrome or mental retardation based on clinical interview
* not participated in DBT treatment during the past year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Deliberate Self-harm Inventory (DSHI; Gratz, 2001) and Lifetime Suicide Attempt Self-Injury interview (LSASI; formerly Lifetime Parasuicide Count, Linehan MM, Comtois KA, unpublished manuscript, 1996) | baseline; 10 weeks; 20 weeks; 3 month follow up
  Self-report measures assessing self-harm and suicidal behaviour

SECONDARY OUTCOMES:
Treatment History Interview (THI-2; Linehan & Heard, 1987) | baseline; 10 weeks; 20 weeks; 3 month follow up
  Assesses for emergency and psychiatric hospitalizations
Barett Impulsiveness Scale (BIS-11; Patton et al., 1995) | Baseline; 10 weeks; 20 weeks; 3 months follow up
  Self-report measure assessing for impulsive behaviour
The State-trait Anger Expression Inventory (STAXI; Spielberger, Krasner & Solomon, 1988) | Baseline; 10 weeks; 20 weeks; 3 months Follow up
  Self-report assessing for anger expressions
The Borderline Evaluation of Severity over time Scale (BEST; Phfolm & Bloom, 1997) | Baseline; 10 weeks; 20 weeks; 3 months Follow up
  self-report measure assessing for severity of BPD symptoms
The Symptom Checklist 90 - Revised (SCL-90-R; Derogatis, 1983) | Baseline; 10 weeks; 20 weeks; 3 months Follow up
  Self-report measure assessing for various psychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Shelley McMain, PhD., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Zeifman RJ, Boritz T, Barnhart R, Labrish C, McMain SF. The independent roles of mindfulness and distress tolerance in treatment outcomes in dialectical behavior therapy skills training. Personal Disord. 2020 May;11(3):181-190. doi: 10.1037/per0000368. Epub 2019 Oct 24. PMID 31647267
- [Derived] Krantz LH, McMain S, Kuo JR. The unique contribution of acceptance without judgment in predicting nonsuicidal self-injury after 20-weeks of dialectical behaviour therapy group skills training. Behav Res Ther. 2018 May;104:44-50. doi: 10.1016/j.brat.2018.02.006. Epub 2018 Mar 1. PMID 29529508
- See also: Related Info — http://www.camh.net/research